CLINICAL TRIAL: NCT07006103
Title: Precision Medicine Applied to Endometrial Cancer (EC)
Brief Title: Precision Medicine Applied to the Study of Endometrial Cancer: Application of NGS for Molecular Classification
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: CEMIC Buenos Aires (Unknown)
Responsible Party: Principal Investigator, Hernan Garcia Rivello, Head of Clinical Pathology Department, Hospital Italiano de Buenos Aires
Other Study IDs: 6760
Record Dates: First submitted 2025-05-16; First posted 2025-06-05 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Cancer, Endometrial Neoplasm
Keywords: endometrial cancer; molecular classification; POLEmut subgroup
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue and DNA extract
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, knowledge about cancer biology has expanded significantly. The study of gene expression profiles has revealed the heterogeneous nature and potential reclassification of the various tumor subtypes based on specific genetic alterations. This is of great importance since it allows a therapeutic approach more directed to the intrinsic characteristics of each tumor (precision medicine).

Integrating clinicopathological information with molecular classification could provide new guidelines when approaching patients with EC, both in preoperative assessment and in adjuvant treatment and surveillance.

The application of molecular classification in endometrial carcinomas shows a subgroup of patients with an excellent prognosis, corresponding to the POLEmut subgroup that could be reclassified with eventual therapeutic de-escalation.

The clinical guidelines for the management of patients with endometrial cancer proposed by ESGO/ESTRO/ESP in 2020 recommend the use of this new classification, and warn that clinical management may be modified by the molecular classification in scenarios where adjuvant chemotherapy is considered (high-grade/high-risk disease).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with a diagnosis of EC diagnosed by histological biopsy and surgically treated sequentially in the participating centers in the last 5 years with clinical follow-up.
* Patients over 18 years of age, diagnosed with CE III-IV by histological biopsy, not susceptible to surgical treatment in each institution during the last 5 years in clinical follow-up. Cases with a diagnosis of carcinosarcoma (a rare subtype of endometrial carcinoma with sarcomatous transdifferentiation) are included.
* Material blocks fixed in formalin and embedded in paraffin with a tumor volume in the paraffin block of at least 1 cm3

Exclusion Criteria:

* The following uterine neoplasms will be excluded:

  * Biphasic tumors (epithelial-mesenchymal) such as adenosarcoma.
  * Mesenchymal neoplasms such as endometrial stromal sarcoma and leiomyosarcomas.
  * Others: primary lymphoproliferative processes of the uterine body; neuroendocrine tumors; Gestational trophoblastic disease, secondary lesions either of the genital tract (example: cervical carcinomas with extension to the endometrium) or of distant sites (breast cancer metastasis).

    * Patients with synchronous endometrial and ovarian carcinoma
    * For technical reasons, they will be excluded
  * tumors smaller than 0.2 cm in which sufficient material cannot be obtained for immunohistochemical and molecular biology determinations.
  * Tumors with severe artifacts due to poor processing, such as autolysis.
  * Samples with low-quality DNA

    * Patients operated on outside participating centers.
    * Patients under 18 years of age.
    * Patients with primary non-surgical treatments (neoadjuvant chemotherapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The endometrium is a female organ
Study Population: Patients of Hospital Italiano de Buenos Aires. Section of Pathological Anatomy, Sequencing and Gynecological Oncology, and the "Norberto Quirno" Center for Medical Education and Clinical Research (CEMIC). Service of Pathological Anatomy, Molecular Pathology, Gynecology, Institute of Oncology, and Institute of Precision Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Distribution of Endometrial Cancer Molecular Subtypes Identified by Immunohistochemistry and POLE Sequencing | At study inclusion (retrospective evaluation of cases from the last 5 years). Units: Percentage of patients per subtype
  Proportion of patients in each of the four molecular subtypes of endometrial cancer (POLE-ultramutated, microsatellite instability hypermutated, copy-number low, copy-number high) determined using immunohistochemistry for MMR proteins and TP53, and NGS-based sequencing of the POLE gene.

SECONDARY OUTCOMES:
Association Between Molecular Subtypes and Histological Risk Categories. | At study inclusion (retrospective evaluation of cases from the last 5 years).
  Proportion of patients with low- versus high-risk histological types within each molecular subtype.
Time to Recurrence by Molecular Subtype | At study inclusion (retrospective evaluation of cases from the last 5 years).
  Time (in months) from diagnosis to first documented relapse, stratified by molecular subtype.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stelloo E, Nout RA, Osse EM, Jurgenliemk-Schulz IJ, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Nijman HW, Putter H, Bosse T, Creutzberg CL, Smit VT. Improved Risk Assessment by Integrating Molecular and Clinicopathological Factors in Early-stage Endometrial Cancer-Combined Analysis of the PORTEC Cohorts. Clin Cancer Res. 2016 Aug 15;22(16):4215-24. doi: 10.1158/1078-0432.CCR-15-2878. Epub 2016 Mar 22. PMID 27006490
- [Background] Talhouk A, McConechy MK, Leung S, Yang W, Lum A, Senz J, Boyd N, Pike J, Anglesio M, Kwon JS, Karnezis AN, Huntsman DG, Gilks CB, McAlpine JN. Confirmation of ProMisE: A simple, genomics-based clinical classifier for endometrial cancer. Cancer. 2017 Mar 1;123(5):802-813. doi: 10.1002/cncr.30496. Epub 2017 Jan 6. PMID 28061006
- [Background] Hoang LN, Kinloch MA, Leo JM, Grondin K, Lee CH, Ewanowich C, Kobel M, Cheng A, Talhouk A, McConechy M, Huntsman DG, McAlpine JN, Soslow RA, Gilks CB. Interobserver Agreement in Endometrial Carcinoma Histotype Diagnosis Varies Depending on The Cancer Genome Atlas (TCGA)-based Molecular Subgroup. Am J Surg Pathol. 2017 Feb;41(2):245-252. doi: 10.1097/PAS.0000000000000764. PMID 28079598
- [Background] Kobel M, Nelson GS. Letter in response to: McAlpine J, Leon-Castillo A, Bosse T. The rise of a novel classification system for endometrial carcinoma; integration of molecular subclasses. J Pathol 2018; 244: 538-549. J Pathol. 2018 Jun;245(2):249-250. doi: 10.1002/path.5068. Epub 2018 Apr 16. No abstract available. PMID 29512840
- [Background] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Background] Bendifallah S, Canlorbe G, Collinet P, Arsene E, Huguet F, Coutant C, Hudry D, Graesslin O, Raimond E, Touboul C, Darai E, Ballester M. Just how accurate are the major risk stratification systems for early-stage endometrial cancer? Br J Cancer. 2015 Mar 3;112(5):793-801. doi: 10.1038/bjc.2015.35. Epub 2015 Feb 12. PMID 25675149
- [Background] Imai K, Kato H, Katayama K, Nakanishi K, Kawano A, Iura A, Konnai K, Onose R, Hirahara F, Miyagi E. A preoperative risk-scoring system to predict lymph node metastasis in endometrial cancer and stratify patients for lymphadenectomy. Gynecol Oncol. 2016 Aug;142(2):273-7. doi: 10.1016/j.ygyno.2016.06.004. Epub 2016 Jun 15. PMID 27268220
- [Background] Bokhman JV. Two pathogenetic types of endometrial carcinoma. Gynecol Oncol. 1983 Feb;15(1):10-7. doi: 10.1016/0090-8258(83)90111-7. PMID 6822361
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338